CLINICAL TRIAL: NCT03958513
Title: Randomized, Double- Blind, Controlled Trial to Evaluate the Effect of Wound Infiltration With Bupivacaine for Post-operative Pain Relief After Laparoscopic Cholecystectomy
Brief Title: To Evaluate the Effect of Wound Infiltration With Bupivacaine for Post-operative Pain Relief After Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Monira Parveen, Principal investigator, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BSMMU/2018/12652
Record Dates: First submitted 2019-05-15; First posted 2019-05-22 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): 0.9% normal saline, 1.5 ml for 1 inch incision, before closure of ports in patients undergoing Laparoscopic Cholecystectomy
  Interventions: Drug: 0.9% normal saline
- Intervention (Experimental): 0.25% Bupivacaine, 1.5 ml per 1 inch incision, before closure of ports in patients undergoing Laparoscopic Cholecystectomy
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — 1.5 ml 0.25% bupivacaine for 1 inch incision will be given before closure of ports in patients undergoing laparoscopic cholecystectomy
  Arms: Intervention
Drug: 0.9% normal saline — 1.5 ml 0.9% NACl for 1 inch incision will be given before closure of ports in patients undergoing laparoscopic cholecystectomy
  Arms: Placebo

SUMMARY:
To evaluate the effect of wound infiltration with 0.25% Bupivacaine in laparoscopic cholecystectomy in terms of pain severity, patient satisfaction level, quality of life, hospital stay and return to job and normal activities.

ELIGIBILITY:
Inclusion criteria

* Patients scheduled to undergo laparoscopic cholecystectomy under general anesthesia at department of surgery and department of hepatobiliary system, BSMMU
* Patients who are eligible according to ASA Ⅰ -Ⅱ
* Female or male, age ≥18 years
* Patients who are scheduled for same anesthetic technique and surgical procedure for laparoscopic cholecystectomy
* Discharge of patient between 12 hour to 36 hour after performing procedure
* Patients given consent for enrollment in study

Exclusion criteria

* Patients known to be allergic to certain recommended drugs
* If patients have history of psychiatric illness
* Patients on chronic analgesic therapy for any other indication
* Patients who are scheduled for different anesthetic technique and surgical procedure for laparoscopic cholecystectomy
* Duration of surgery more than 1 hour
* Patients undergoing laparoscopic cholecystectomy for complex gallbladder disease such as incidental gallbladder pancreatitis, gallstone pancreatitis, cholecystoduodenal fistula, mirizzi syndrome
* Special population group such as children, pregnant woman, patients with cirrhosis, diabetics
* Duration of operative procedure more than 1 hour

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Post-operative pain: VAS | 12 hours
  Post-operative pain in visual analog scale ranging 0 to100
Post-operative pain: rating scale | 12 HOURS
  Post-operative pain in numerical rating scale ranging 0 to 4

SECONDARY OUTCOMES:
Patient Satisfaction Level: questionnaire | 24 hour
  Patient Satisfaction Level is measured with revised american pain society outcome questionnaire. 12 questions are present.
Hospital stay | 3-5 days
  Time frame for hospital discharge
Pain during hospital discharge: VAS | 3-5days
  visual analog scale score during hospital discharge rangibg 0-100
Time taken to return to job and normal activities | 15-30 days
Assesment of quality of life: index | 15th and 30th post-operative day
  Quality of life is measured with gastrointestinal quality of life index. there are 36 questions . it will measure quality of life after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No